CLINICAL TRIAL: NCT04250792
Title: Efficacy of Low Dose Naltrexone in Psoriasis; Clinical Trial in a Tertiary Care Hospital of Karachi.
Brief Title: Efficacy of Low Dose Naltrexone in Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Sidra Khan, Principal investigator, Jinnah Postgraduate Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO.F.2-81/2018-GENL/9009/JPMC
Record Dates: First submitted 2020-01-26; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Psoriasis
Keywords: Low dose naltrexone; psoriasis; Psoriasis area severity index
MeSH Terms: conditions — Psoriasis | interventions — Naltrexone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Low dose naltrexone was prescribed to the patients affected with psoriasis.
  Interventions: Drug: Naltrexone Pill

INTERVENTIONS:
Drug: Naltrexone Pill — role of low dose naltrexone in patients affected with psoriasis
  Other Names: low dose naltrexone

SUMMARY:
Objective of the study is to determine the efficacy of low dose naltrexone in the patients of psoriasis, which is a chronic relapsing and remitting disease. A non-randomized clinical trial was carried out in the Department of dermatology in Jinnah Postgraduate Medical Center, Karachi. All patients with mild, moderate and severe psoriasis with age above 13 years without any co-morbid, were prescribed tablet Naltrexone 6 mg daily after assessing PASI, BSA and DLQI scores before starting treatment. Patients were called monthly for follow up to monitor lipid profiles and liver function tests. After 3 months of treatment, PASI, BSA and DLQI scores were assessed again. The results were significant when analysed with paired t test in SPSS 23.

DETAILED DESCRIPTION:
Psoriasis is a chronic T-cell mediated disorder. The activated T cell secretes cytokines that result in keratinocytes hyper-proliferation and abnormal differentiation. These cytokines result in chemo-taxis of neutrophils and lymphocytes in skin. It is a multi-factorial disease. Individual has genetic susceptibility for psoriasis, but environmental factors trigger the disease like infections, drugs, cold, trauma and stress. It is a multi-system disease but mainly affects skin, nails and joints. It impacts adversely on patients' quality of life, causes embarrassment, limitation in clothing choice, psychological distress which further aggravates the disease. It impacts economically due to off days from work as well. In its most common form, it presents as salmon pink plaques, covering with thick silver scales, mostly on scalp, trunk, buttocks and external surfaces of limbs.

In the management of psoriasis, there are multiple treatment options which includes topical, systemic and photo-therapy. But all have their side effects and contraindication. Low dose naltrexone(LDN) is an attractive emergent therapy with analgesic, anti-pruritic and anti-inflammatory properties for various dermatological disorders including psoriasis. In this study, the effectiveness of low dose naltrexone in cases of psoriasis was assessed.

The study was conducted in the department of dermatology in Jinnah Postgraduate Medical Centre, Karachi, after receiving approval letter from the institutional ethical and research committee of the hospital.Forty two patients were selected of either gender with age ranging from 13-60 years, after excluding hypertension, cardiovascular disorders, pregnancy and lactation. The procedure has been explained to each patient & written consent has been taken. Before prescribing LDN treatment, Psoriasis area and severity index(PASI), Body surface area(BSA) and Dermatology life quality index(DLQI) has been calculated. Each case has prescribed tablet naltrexone 6mg daily after checking all baselines investigations of complete blood picture , renal and liver function profiles. The cases were asked to follow up monthly to observe patient compliance, response of medicine and its side effects. After 3 months of treatment, PASI, BSA and DLQI have been calculated to assess the effectiveness of treatment.

PASI score is used to measure the severity and extent of disease, in terms of intensities of erythema, induration and scaling of lesion and the area of body involved with disease.

Body surface area (BSA) is calculated through 'rule of nine' which is a convenient and rapid method of estimating the extent of body surface area affected with disease. If BSA is <3%, 3-10%, or >10%, it is categorized as mild, moderate and severe disease, respectively.

The dermatology life quality index is a simple questionnaire, that consists of 10 questions to assess the impact of disease and its treatment on daily activities and the impact on the social behavior of the patients. DLQI scores has been interpreted in terms of effect of disease on patients' life as follows:

* 0-1 = No effect
* 2-5 = Small effect
* 6-10 = Moderate effect
* 11-20 = Very large effect
* 21-30 = Extremely large effect After 3 months, all three scores were assessed again to observe the effectiveness of treatment. The evaluation was done by SPSS version 23. The side effects were assessed regarding nausea, headache, decreased appetite, dizziness, palpitation, liver enzymes level, renal and complete blood profiles.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 13 years
* maximum age 60 years
* both males and females affected with mild, moderate and severe psoriasis.

Exclusion Criteria:

* hypertension
* cardiovascular disorders
* pregnancy
* lactation
* renal failure
* liver failure
* hypersensitivity to drug

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
change in the severity of disease | 12 weeks.
  change in the percentage of area of body involved with disease (1 hand = 1%)

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ghafoor, FCPS, Study Director — Jinnah postgraduate medical centre, Karachi
Locations (1):
- Jinnah postgraduate medical centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rendon A, Schakel K. Psoriasis Pathogenesis and Treatment. Int J Mol Sci. 2019 Mar 23;20(6):1475. doi: 10.3390/ijms20061475. PMID 30909615
- [Background] Zashin S. Sjogren's Syndrome: Clinical Benefits of Low-dose Naltrexone Therapy. Cureus. 2019 Mar 11;11(3):e4225. doi: 10.7759/cureus.4225. PMID 31123647
- [Result] Beltran Monasterio EP. Low-dose Naltrexone: An Alternative Treatment for Erythrodermic Psoriasis. Cureus. 2019 Jan 23;11(1):e3943. doi: 10.7759/cureus.3943. PMID 30937241